CLINICAL TRIAL: NCT01127061
Title: A Randomized Trial of Moderate Intensity Exercise Training in Hypertrophic Cardiomyopathy
Brief Title: Study of Exercise Training in Hypertrophic Cardiomyopathy
Acronym: RESET-HCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Sara Saberi, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RESET-HCM
Record Dates: First submitted 2010-05-17; First posted 2010-05-20 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Cardiomyopathy, Hypertrophic
Keywords: Hypertrophic Cardiomyopathy; Exercise; Oxygen consumption
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator who randomized participants was blinded to participant PHI. Investigators who interpreted all data and assessed outcomes were masked to randomization status.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Training (Experimental): Participants in the exercise group will undergo 4 months of training, 4-7 days per week with a minimum of 20 minutes per day. The protocol will be custom designed in consultation with an exercise physiologist based on data from the initial cardiopulmonary stress test. Exercise regimen will begin at a low level of intensity then increase in duration and training intensity to a goal of 60 minutes a day and 70% of the heart rate reserve during the 1st month of the study protocol with maintenance of the program thereafter. There is no need to come to a participating site for actually doing the exercise regimen. No strength training or burst activity will be prescribed and all activities will fall well within the recommended national guidelines for recreational exercise.
  Interventions: Behavioral: Exercise training
- Usual Activity (No Intervention): Participants in this group are not restricted in their activities. They simply are not guided in their physical activities by the study team. At the end of the 4 month study period, they will also receive an individualized exercise prescription for personal use.

INTERVENTIONS:
Behavioral: Exercise training — 4 months of exercise training that is custom-designed based on individual cardiopulmonary stress test data. Regimen starts at low intensity (60% of heart rate reserve) and frequency (20 minutes, 3 days per week) and increases with a goal of 70% of heart rate reserve and exercising 60 minutes 4-7 days per week.
  Arms: Exercise Training

SUMMARY:
The investigators propose a pilot randomized controlled trial to determine the safety and potential benefits of moderate intensity exercise in patients with hypertrophic cardiomyopathy. The investigators hypotheses are that exercise parameters derived from a baseline cardiopulmonary exercise test will target an appropriately safe level of exercise intensity that will not cause significant arrhythmias or exacerbate symptoms and that exercise training for 4 months will result in significant improvements in peak oxygen consumption (peak VO2) and quality of life, with neutral effects on the clinical characteristics.

DETAILED DESCRIPTION:
The goal of this randomized clinical pilot trial is to establish the safety profile and potential benefits of moderate intensity exercise in patients with hypertrophic cardiomyopathy (HCM). Participation in competitive athletics is associated with an increased risk of sudden cardiac death (SCD) in individuals with structural heart disease, including HCM. This has appropriately led to the establishment of national guidelines based on expert opinion that discourage participation in high intensity competitive sports, burst exertion (e.g., sprinting), or isometric exercise (e.g., heavy lifting). Non-competitive, low to moderate intensity exercise is allowable, although many physicians and HCM patients are still understandably apprehensive. Data on the safety of a recreational exercise program, and how to gauge appropriate intensity level, are desperately needed so that HCM patients can reap the well established health benefits of regular physical activity. Limited, but compelling animal data suggest that moderate intensity exercise is not only safe, but may also prevent or even reverse cardiac hypertrophy, fibrosis, myocellular disarray, and apoptosis associated with HCM. There are no published studies on exercise in patients with HCM, although large clinical trials in heart failure have shown exercise training to be safe, to improve peak VO2 and quality of life, and to lower cardiovascular mortality. The pilot randomized control trial proposed here is the first to determine the safety of moderate intensity exercise training and explore its potential benefits in patients with HCM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 80.
* Diagnosis of HCM, defined by the presence of unexplained left-ventricular hypertrophy > 13 mm in any wall segment.
* Agreement to be a participant in the study protocol and willing/able to return for follow-up.

Exclusion Criteria:

* History of exercise-induced syncope or arrhythmias (ventricular tachycardia or non-sustained ventricular tachycardia).
* Medically refractory left ventricular outflow tract obstruction being evaluated for septal reduction therapy.
* Less than 3 months post septal reduction therapy (surgery or catheter based intervention).
* Hypotensive response to exercise (> 20 mm Hg drop in systolic blood pressure from peak blood pressure to post exercise blood pressure).
* Pregnancy.
* Implantable Cardioverter-Defibrillator (ICD) placement in last 3 months or scheduled.
* Left ventricular systolic dysfunction (left ventricular ejection fraction < 55% by echocardiography).
* Worsening clinical status in the last 3 months, advanced heart failure (New York Heart Association class IV symptoms) or angina (Canadian Cardiovascular Society class IV symptoms).
* Life expectancy less than 12 months.
* Inability to exercise due to orthopedic or other non-cardiovascular limitations.
* Unwillingness to refrain from competitive sports, burst activity, or heavy isometric exercise for the duration of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Saberi, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Michigan Cardiovascular Center, Ann Arbor, Michigan

REFERENCES:
- [Derived] Saberi S, Wheeler M, Bragg-Gresham J, Hornsby W, Agarwal PP, Attili A, Concannon M, Dries AM, Shmargad Y, Salisbury H, Kumar S, Herrera JJ, Myers J, Helms AS, Ashley EA, Day SM. Effect of Moderate-Intensity Exercise Training on Peak Oxygen Consumption in Patients With Hypertrophic Cardiomyopathy: A Randomized Clinical Trial. JAMA. 2017 Apr 4;317(13):1349-1357. doi: 10.1001/jama.2017.2503. PMID 28306757

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise Training: Participants in the exercise group will be follow an individualized moderate-intensity exercise prescription (designed in consultation with an exercise physiologist based on data from the initial cardiopulmonary stress test). Exercise regimen will begin at a low level of intensity (3 sessions per week, 20 minutes per session, at a heart rate corresponding to 60% of heart rate reserve), then increase in duration and training intensity to a goal of up to 60 minutes per session, 4 to 7 sessions per week, at 70% of the heart rate reserve during the 1st month of the study protocol with maintenance of the program thereafter. No strength training or burst activity will be prescribed and all activities will fall well within the recommended national guidelines for recreational exercise.
Period: Overall Study
Arm/Group | Exercise Training | Usual Activity
Started | 67 | 69
Completed | 57 | 56
Not Completed | 10 | 13
Not completed — Lost to Follow-up | 7 | 10
Not completed — Physician Decision | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Usual Activity: Participants in this group are not restricted in their activities. They simply are not guided in their physical activities by the study team. At the end of the 4-month study period, they will also receive an individualized exercise prescription for personal use.
- Total: Total of all reporting groups
Arm/Group | Exercise Training | Usual Activity | Total
Number analyzed (Participants) | 67 | 69 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (13.2) | 50.0 (13.5) | 50.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 38 | 41 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 63 | 67 | 130
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 56 | 63 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 67 | 69 | 136
Weight, Continous [Mean (Standard Deviation); unit: kg] | 90.5 (18.3) | 92.6 (15.7) | 91.6 (17.0)
Peak oxygen consumption (VO2), Continuous [Mean (Standard Deviation); unit: mL/kg/min] | 21.3 (6.3) | 22.5 (7.2) | 21.9 (6.8)
Maximal left ventricular wall thickness [Mean (Standard Deviation); unit: mm] — As measured by echocardiography
  mm | 21 (5) | 21 (6) | 21 (5.9)
Left ventricular outflow tract obstruction at rest [Count of Participants; unit: Participants] — Defined as resting left ventricular outflow tract peak pressure gradient 30 mm Hg or greater.
  Participants | 11 | 12 | 23
Peak left ventricular pressure gradient at rest [Mean (Standard Deviation); unit: mm Hg] | 15.2 (14) | 20.7 (27.2) | 18.0 (21.8)
Peak left ventricular outflow gradient with Valsalva maneuver [Mean (Standard Deviation); unit: mm Hg] — Population: Data was not obtained or was not reliably measured in every study participant.
  mm Hg
    number analyzed (Participants) | 60 | 60 | 120
    (all) | 23.6 (24.6) | 31.8 (37.3) | 27.7 (31.7)
Peak left ventricular outflow gradient after exercise [Mean (Standard Deviation); unit: mm Hg] — Population: Data was not obtained or was not reliably measured in every study participant.
  mm Hg
    number analyzed (Participants) | 66 | 68 | 134
    (all) | 48.1 (43.5) | 57.0 (51.9) | 52.6 (47.4)
Left atrial volume index [Mean (Standard Deviation); unit: mL/m2] | 47.4 (15.6) | 46.1 (14.3) | 46.7 (14.9)
Left ventricular ejection fraction [Mean (Standard Deviation); unit: %] | 70.6 (4.0) | 70.8 (4.3) | 70.7 (4.1)
Total delayed gadolinium enhancement mass [Mean (Standard Deviation); unit: g] — As measured by cardiac magnetic resonance imaging Population: Cardiac magnetic resonance imaging was not obtained in every participant due to presence of implantable cardioverter-defibrillator, permanent pacemaker, or claustrophobia.
  g
    number analyzed (Participants) | 28 | 30 | 58
    (all) | 4.7 (6.7) | 4.9 (10.3) | 4.8 (8.7)
New York Heart Association Class II-III [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification system is used to classify severity of heart failure symptoms as follows with Class I indicating best outcome and Class IV, the worst:
  Class I: No limitation of physical activity.
  Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in symptoms (fatigue, palpitations, or shortness of breath).
  Class III: Comfortable at rest. Less than ordinary physical activity results in symptoms.
  Class IV: Symptoms of heart failure at rest.
  Participants | 23 | 23 | 46
B-type natriuretic peptide [Median (Inter-Quartile Range); unit: pg/mL] | 79 [27 to 186] | 83 [38 to 200] | 79 [31 to 192]
History of implantable cardioverter defibrillator [Count of Participants; unit: Participants] | 25 | 21 | 46
History of ventricular tachycardia, ventricular fibrillation, or sudden cardiac death [Count of Participants; unit: Participants] | 3 | 2 | 5
History of nonsustained ventricular tachycardia [Count of Participants; unit: Participants] | 9 | 10 | 19
History of atrial fibrillation or flutter [Count of Participants; unit: Participants] | 14 | 8 | 22
History of septal reduction procedure [Count of Participants; unit: Participants] | 20 | 15 | 35
History of hypertension [Count of Participants; unit: Participants] | 14 | 16 | 30
Beta-blocker use [Count of Participants; unit: Participants] | 41 | 51 | 92
Calcium channel blocker use [Count of Participants; unit: Participants] | 15 | 14 | 29
Sarcomere mutation [Count of Participants; unit: Participants]
  No testing | 5 | 1 | 6
  Pathogenic | 33 | 25 | 58
  Variant of uncertain significance | 8 | 6 | 14
  Negative | 21 | 37 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Oxygen Consumption (Peak VO2)
Description: Cardiopulmonary exercise testing was performed at study enrollment and termination (4 months apart). Peak VO2 was measured at each time point in each subject and change in peak VO2 over time was calculated. The change in Peak VO2 was compared between the study arms.
Time Frame: At study Enrollment and 4 months later
Population: These numbers reflect the attrition rates seen in the study.
Measure: Mean (95% Confidence Interval); unit: mL/kg/min
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 57 | 56
mL/kg/min | 1.35 [0.50 to 2.21] | 0.08 [-0.62 to 0.79]

2. Other Pre Specified Outcome: Change in Quality of Life
Description: Quality of life (QOL) questionnaires (Minnesota Living With Heart Failure Questionnaire, MLHF; Quick Inventory of Depressive Symptomatology-Self Report, QIDS-SR16; and the 36-Item Short-Form Health Survey Version 2, SF-36v2) were administered at study enrollment and termination (4 months later). Change over time was compared between study arms.
  MLHF: range, 0-105; higher scores indicate worse QOL QIDS-SR16: range, 0-27; higher scores indicate more severe depression SF-36v2: 8 subscales and 2 component summary scores; range, 1-100; lower scores indicate more disability; minimal clinically important difference, 3 to 5 points
Time Frame: At study enrollment and 4 months later
Population: These numbers reflect attrition rates in the study.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 57 | 56
units on a scale
  Change in Physical Functioning Scale, SF-36v2: number analyzed (Participants) | 51 | 50
  Change in Physical Functioning Scale, SF-36v2 | 5.7 [1.6 to 9.8] | -2.5 [-6.2 to 1.3]
  Change in Role Physical Scale, SF-36v2: number analyzed (Participants) | 51 | 49
  Change in Role Physical Scale, SF-36v2 | 0.1 [-0.5 to 0.8] | -0.04 [-1.7 to 1.6]
  Change in Bodily Pain Scale, SF-36v2: number analyzed (Participants) | 51 | 49
  Change in Bodily Pain Scale, SF-36v2 | 1.1 [-3.4 to 5.8] | -2.2 [-8.3 to 3.9]
  Change in General Health Perception Scale, SF-36v2: number analyzed (Participants) | 51 | 50
  Change in General Health Perception Scale, SF-36v2 | 4.1 [0.03 to 8.2] | 0.2 [-4.3 to 4.6]
  Change in Energy/Fatigue Scale, SF-36v2: number analyzed (Participants) | 50 | 48
  Change in Energy/Fatigue Scale, SF-36v2 | 3.5 [-0.9 to 7.9] | 6.0 [1.5 to 10.5]
  Change in Social Functioning Scale, SF-36v2: number analyzed (Participants) | 51 | 50
  Change in Social Functioning Scale, SF-36v2 | 1.0 [-3.3 to 5.3] | 3.0 [-3.0 to 8.9]
  Change in Role Emotional Scale, SF-36v2: number analyzed (Participants) | 51 | 49
  Change in Role Emotional Scale, SF-36v2 | 0 [0 to 0] | 0.5 [-0.1 to 1.1]
  Change in Emotional Well-Being Scale, SF-36v2: number analyzed (Participants) | 50 | 48
  Change in Emotional Well-Being Scale, SF-36v2 | 2.8 [-1.5 to 7.0] | 4.5 [0.7 to 8.3]
  Change in Physical Component Summary, SF-36v2: number analyzed (Participants) | 50 | 47
  Change in Physical Component Summary, SF-36v2 | 1.3 [0.2 to 2.3] | -0.1 [-1.4 to 1.2]
  Change in Mental Component Summary, SF-36v2: number analyzed (Participants) | 50 | 47
  Change in Mental Component Summary, SF-36v2 | 1.3 [-0.3 to 2.8] | 1.9 [0.4 to 3.4]
  Change in QIDS-SR16 | -0.9 [-1.7 to -0.1] | -0.8 [-1.7 to 0.1]
  Change in MLHF Total Score: number analyzed (Participants) | 54 | 54
  Change in MLHF Total Score | -3.4 [-6.6 to -0.2] | -2.4 [-6.1 to 1.4]
  Change in Physical Dimension, MLHF: number analyzed (Participants) | 55 | 55
  Change in Physical Dimension, MLHF | -1.1 [-2.8 to 0.7] | -0.2 [-1.8 to 1.3]
  Change in Emotional Dimension, MLHF: number analyzed (Participants) | 56 | 55
  Change in Emotional Dimension, MLHF | -0.9 [-2.0 to 0.2] | -2.1 [-3.5 to -0.6]

3. Other Pre Specified Outcome: Change in Concentration of Brain Natriuretic Peptide (BNP)
Description: Blood will be drawn to evaluate BNP at study enrollment and termination (4 months later). Change over time was compared between study arms.
Time Frame: At study enrollment and 4 months later
Population: These numbers reflect attrition rates in the study, as well as, whether data was obtained at each time point.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 44 | 44
pg/mL | 5 [-10 to 27] | 9 [-14 to 40]

4. Other Pre Specified Outcome: Change in Scar Volume
Description: Cardiac MRI was performed in all patients without implantable devices/claustrophobia requiring sedation at study enrollment and termination (4 months later). Scar volume was calculated as total delayed gadolinium enhancement mass at each time interval. Change over time was compared between study arms.
Time Frame: At study enrollment and 4 months later
Population: These numbers reflect attrition rates in the study, as well as, whether cardiac MRI was performed.
Measure: Mean (95% Confidence Interval); unit: g
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 29 | 30
g | 0.35 [-0.2 to 0.9] | -0.03 [-0.7 to 0.7]

5. Other Pre Specified Outcome: Change in Systolic Function as Measured by Left Ventricular Ejection Fraction.
Description: Echocardiography was performed at study enrollment and termination. Left ventricular ejection fraction was visually estimated on each echocardiogram. Change over time was compared by study arm assignment.
Time Frame: At study enrollment and 4 months later
Population: These numbers reflect attrition rates in the study, as well as, whether data was reliably obtained at each time point.
Measure: Mean (95% Confidence Interval); unit: percentage of ventricular blood
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 55 | 58
percentage of ventricular blood | -0.2 [-0.9 to 0.4] | -0.2 [-1.3 to 1.0]

6. Other Pre Specified Outcome: Change in Degree of Left Ventricular Outflow (LVOT) Obstruction.
Description: Cardiopulmonary exercise testing in combination with echocardiography was performed at study enrollment and termination (4 months). Peak left ventricular outflow gradients were obtained at rest, with Valsalva and after exercise at each time point. The change over time was compared by study arm assignment.
Time Frame: At study enrollment and 4 months later
Population: These numbers reflect the rate of attrition in the study, as well as, whether data was reliably obtained at each time point.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 55 | 58
mm Hg
  Change in peak LVOT gradient at rest | 4.2 [-1.5 to 9.9] | -3.8 [-9.2 to 1.5]
  Change in peak LVOT gradient with Valsalva | 9.6 [-1.5 to 9.9] | -3.0 [-13.0 to 7.0]
  Change in peak LVOT gradient after exercise | 3.3 [-4.8 to 11.4] | -4.2 [-13.9 to 5.5]

7. Other Pre Specified Outcome: Change in Maximal Left Ventricle Wall Thickness
Description: Magnitude or distribution of cardiac hypertrophy or left ventricular dimensions were a pre-specified outcome. Maximal left ventricle (LV) wall thickness (mm) was measured by cardiac MRI performed at study enrollment and termination (4 months later) and change over time was compared between study arms. Cardiac MRI was only be performed in those who do not have implantable devices or claustrophobia significant enough to require sedation.
Time Frame: At study enrollment and 4 months later
Population: These numbers reflect the number of participants that underwent cardiac MRI and attrition rates in the study.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 30 | 31
mm | -0.3 [-0.9 to 0.2] | -0.6 [-1.1 to -0.1]

8. Other Pre Specified Outcome: Change in Diastolic Function
Description: Diastolic function was assessed at each time point and categorized as indeterminate diastolic function, grade I diastolic dysfunction and grade II-III diastolic dysfunction, according to American Society of Echocardiography criteria. Number of participants whose findings fell into each category was calculated and % change over time was compared between study arms. Indeterminate indicates diastolic function could not be accurately categorized. Grade I diastolic dysfunction indicates least severe in terms of outcome measure and Grade III, most severe.
Time Frame: At study Enrollment and 4 months later
Population: These numbers reflect attrition rates in the study, as well as, whether data was reliably obtained at each time point.
Measure: Mean (95% Confidence Interval); unit: % of participants
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 54 | 58
% of participants
  Change in % Indeterminate diastolic dysfunction | 16.4 [6.4 to 26.5] | 15.9 [7.1 to 24.8]
  Change in % Grade I diastolic dysfunction | -11.9 [-24.3 to 0.5] | -13.0 [-26.0 to -0.1]
  Cahnge in % Grade II-III diastolic dysfunction | 0 [-11.9 to 11.9] | 1.7 [-10.8 to 14.3]

9. Other Pre Specified Outcome: Change in Left Ventricular Mass Index
Description: Magnitude or distribution of cardiac hypertrophy or left ventricular dimensions were a pre-specified outcome. Left ventricular mass index was measured by cardiac MRI at study enrollment and termination (4 months later) and change over time was compared between study arms. Cardiac MRI was only be performed in those who do not have implantable devices or claustrophobia significant enough to require sedation.
Time Frame: At study enrollment and 4 months later
Population: These numbers reflect the number of participants who were able to undergo cardiac MRI and attrition rates in the study.
Measure: Mean (95% Confidence Interval); unit: g/m2
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 28 | 29
g/m2 | 2.8 [-0.8 to 6.3] | 0.7 [-1.4 to 2.9]

10. Other Pre Specified Outcome: Change in Left Ventricular End Diastolic Volume Index
Description: Magnitude or distribution of cardiac hypertrophy or left ventricular dimensions were a pre-specified outcome. Left ventricular end diastolic volume index was measured by cardiac MRI at study enrollment and termination (4 months later) and change over time was compared between study arms. Cardiac MRI was only be performed in those who do not have implantable devices or claustrophobia significant enough to require sedation.
Time Frame: At study enrollment and 4 months later
Population: These numbers reflect the number of participants who were able to undergo cardiac MRI and attrition rates in the study.
Measure: Mean (95% Confidence Interval); unit: mL/m2
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 28 | 30
mL/m2 | 1.1 [-2.3 to 4.5] | 0.5 [-2.1 to 3.2]

11. Other Pre Specified Outcome: Change in Left Ventricular End Systolic Volume Index
Description: Magnitude or distribution of cardiac hypertrophy or left ventricular dimensions were a pre-specified outcome. Left ventricular end systolic index was measured by cardiac MRI at study enrollment and termination (4 months later) and change over time was compared between study arms. Cardiac MRI was only be performed in those who do not have implantable devices or claustrophobia significant enough to require sedation.
Time Frame: At study enrollment and 4 months later
Population: These numbers reflect number of participants who were able to undergo cardiac MRI and attrition rates in the study.
Measure: Mean (95% Confidence Interval); unit: mL/m2
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 28 | 30
mL/m2 | 0.4 [-1.4 to 2.2] | -0.1 [-2.4 to 2.1]

12. Other Pre Specified Outcome: Change in Left Atrial Size
Description: Magnitude or distribution of cardiac hypertrophy or left ventricular dimensions were a pre-specified outcome. Left atrial size was measured by echocardiography at study enrollment and termination (4 months later) and change over time was compared between study arms.
Time Frame: At study enrollment and 4 months later
Population: These numbers reflect the attrition rates in the study as well as ability to accurately obtain the data given image quality.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 54 | 58
mm | 0.9 [-0.7 to 2.4] | -0.1 [-0.9 to 0.8]

13. Other Pre Specified Outcome: Change in Left Atrial Volume Index
Description: Magnitude or distribution of cardiac hypertrophy or left ventricular dimensions were a pre-specified outcome. Left atrial volume index was measured by echocardiography at study enrollment and termination (4 months later) and change over time was compared between study arms.
Time Frame: At study enrollment and 4 months later
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: mL/m2
Arm/Group | Exercise Training | Usual Activity
Number analyzed (Participants) | 55 | 55
mL/m2 | -1.0 [-4.1 to 2.0] | 0.7 [-2.9 to 4.3]

ADVERSE EVENTS:
Arm/Group | Exercise Training | Usual Activity
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/69
Other Adverse Events (participants affected / at risk) | 34/67 | 38/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exercise Training (N=67) | Usual Activity (N=69)
Nonsustained ventricular tachycardia (Cardiac disorders) | 19 | 15 — Number of participants in each group with arrhythmia detected on 24-hour continuous rhythm monitoring on enrollment or at end or study or during automatically triggered arrhythmia detection monitoring in the first month of the study participation.
Atrial fibrillation (Cardiac disorders) | 5 | 7 — Number of participants in each group with arrhythmia detected on 24-hour continuous rhythm monitoring on enrollment or at end or study or during automatically triggered arrhythmia detection monitoring in the first month of the study participation.
Supraventricular tachycardia (Cardiac disorders) | 23 | 29 — Number of participants in each group with arrhythmia detected on 24-hour continuous rhythm monitoring on enrollment or at end or study or during automatically triggered arrhythmia detection monitoring in the first month of the study participation.
Syncope (Cardiac disorders) | 0 | 2
Major musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 3 | 2 — Number of participants in each group with a major injury with associated persistent incapacity
Minor musculoskeletal injury (Metabolism and nutrition disorders) | 0 | 1 — Number of participants in each group with a minor injury with associated mild or moderate discomfort

LIMITATIONS AND CAVEATS:
Potential for sampling bias. Modest effect size of exercise training. Not powered to assess safety. Not possible to blind patients to treatment assignment. Prescription only incorporated moderate-intensity aerobic exercise in adult patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No